CLINICAL TRIAL: NCT01860157
Title: A Randomized Controlled Study of H1-Coil rTMS for Treatment-Resistant Late-Life Depression
Brief Title: Deep rTMS for Treatment-Resistant Late-life Depression
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Brainsway (Industry)
Responsible Party: Principal Investigator, Daniel Blumberger, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 107/2011
Record Dates: First submitted 2013-05-18; First posted 2013-05-22 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Major Depressive Disorder
Keywords: rTMS; depression; magnetic
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham H1 Coil (Sham Comparator): deep rTMS sham treatment
  Interventions: Device: Brainsway H1-Coil Deep TMS System (Sham treatment)
- Active H1 (Active Comparator): deep rTMS active treatment
  Interventions: Device: Brainsway H1-Coil Deep TMS System

INTERVENTIONS:
Device: Brainsway H1-Coil Deep TMS System (Sham treatment) — In the sham treatment,the electrical field induced by the sham coil cannot invoke any action potentials and if no action potentials are induced, then the electric field is insignificant and there is no treatment effect on the brain.
  Arms: Sham H1 Coil
Device: Brainsway H1-Coil Deep TMS System — Deep Transcranial Magnetic Stimulation (DTMS) is a new form of TMS which allows direct stimulation of deeper neuronal pathways than the standard TMS. The H-coil is a novel DTMS coil designed to allow deeper brain stimulation without a significant increase of electric fields induced in superficial cortical regions
  Arms: Active H1

SUMMARY:
In this study, the investigators will be examining the effects of the deep repetitive transcranial magnetic stimulation (rTMS) using the H1 coil in patients over the age of 60 who have been unable to tolerate or failed to respond to antidepressant medications. The coil was designed to stimulate deeper regions of the left DLPFC. The investigators propose that active stimulation with the H1 coil will result in higher remission rates than placebo stimulation but will have a similar tolerability and safety profile.

DETAILED DESCRIPTION:
This study is a randomized double blind, sham controlled study to evaluate the safety and efficacy of H1-coil rTMS as a treatment for patients over 60 years of age with major depressive disorder who have not tolerated or failed to respond to antidepressant medications. The study duration is 4-6 weeks in length. The acute phase is 4 weeks of 5 daily treatments followed by 2 weeks of biweekly treatment if remission is achieved at the 4 week mark. Symptom change and remission criteria will be assessed using the HRDS-24 item. Cognition will be assessed using a validated battery.

ELIGIBILITY:
Inclusion Criteria:

* outpatients
* voluntary and competent to consent to treatment
* SCID for DSM-IV confirmed diagnosis of major depressive disorder, single or recurrent
* between the ages of 60 and 85
* failed to achieve a clinical response to an adequate dose of an antidepressant based on an ATHF score of ≥ 3 in the current episode OR have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF 1 or 2)
* a score of ≥ 22 on the HDRS-24
* no increase or initiation of any psychotropic medication in the 4 weeks prior to screening
* able to adhere to the treatment schedule
* pass the TMS safety screening questionnaire
* have normal thyroid functioning based on pre-study blood work

Exclusion Criteria:

* history of DSM-IV substance dependence or abuse within the last 3 months
* concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
* acutely suicidal
* pregnant
* lifetime SCID diagnosis of Bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
* SCID diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder) assessed by a study investigator to be primary and causing greater impairment than MDD
* SCID diagnosis of any personality disorder and assessed by a study investigator to be primary and causing greater impairment than MDD
* have presumed or probably dementia, as defined by Mini Mental Status Exam (MMSE)<26 and clinical evidence of dementia
* failed a course of ECT within the current depressive episode
* a significant neurological disorder or insult, including, but no limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
* on a dose of Buprioprion greater than 300mg per day
* have an intracranial implant(e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
* if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions , or the therapeutic focus over the duration of the study
* clinically significant laboratory abnormality, in the opinion of the investigator
* currently (or in the last 4 weeks) take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy
* inability to communicate in English
* non-correctable clinically significant sensory impairment (i.e cannot hear well enough to cooperate with interview)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-06; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HDRS-24 | 4 weeks
  Remission defined as HDRS-24 </= 10

SECONDARY OUTCOMES:
Mean change in HDRS-24 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Blumberger, MD, FRCPC, Principal Investigator — Centre for Addiction and Mental Health; Zafiris J Daskalakis, Md, FRCPC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada